CLINICAL TRIAL: NCT01668628
Title: Quality of Life and Depression in Peritoneal Dialysis Patients and Hemodialysis Patients
Brief Title: Quality of Life and Depression in Dialysis Patients
Acronym: QOLD
Status: Completed | Type: Observational
Sponsor: Fresenius Medical Care Korea (Industry)
Responsible Party: Sponsor
Other Study IDs: QOLD_01_052012
Record Dates: First submitted 2012-05-24; First posted 2012-08-20 (Estimated); Results first posted 2015-09-24 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-08

CONDITIONS: Chronic Kidney Disease Stage 5
Keywords: quality of life; depression; BCM (body composition minitor); hydrational status
MeSH Terms: conditions — Renal Insufficiency, Chronic; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Incident PD patients: First treatment for end stage of renal disease (ESRD) by any peritoneal dialysis modality within 30 days prior to or following enrollment (patients may be enrolled prior to commencing first treatment if there is clear indication that the treatment modality is continuous ambulatory peritoneal dialysis (CAPD) or automated peritoneal dilaysis (APD) and they consent in advance to enter the study) and patients who don't have any experience of dialysis treatment before this study
- Prevalent PD patients: Prevalent peritoneal dialysis(PD) patients who are under peritoneal dialysis treatment more than 6 months
- Prevalent HD patients: Prevalent hemodialysis(HD) patients who are under hemodialysis treatment more than 6 months

SUMMARY:
The aim of this study is to evaluate quality of life (QOL) and depression in peritoneal dialysis patients compare to hemodialysis patients and assess hydration effect on QOL and depression over time.

DETAILED DESCRIPTION:
In dialysis patients, low QOL and depression affects clinical outcomes such as morbidity and mortality.

Therefore at the point of treating dialysis patients, It is important to provide not only physical health but also psychosocial health.

QOL could be decided by physical health (i.e. sign and symptom, laboratory results, death) and psychological health (i.e. fatigue, pain, consciousness of health and satisfaction).

And also generally it is well known that physical and psychological functions in dialysis patients are decreased.

And especially depression is common disease in dialysis patients. It is also well known that about from 25 to 50 percent of dialysis patients have depression which could result in low QOL moreover hospitalization, complication, and mortality.

But there is no QOL and depression study with hydration status. Therefore the investigators would like to explore it.

The objective of the study is to evaluate quality of life (QOL) and depression in dialysis patients and assess the hydration effect on QOL and depression over time

ELIGIBILITY:
Inclusion Criteria:

* Dialysis patients, age from 18 years to 75 years
* Incident continuous ambulatory peritoneal dialysis(CAPD) or automated peritoneal dialysis(APD) patients who don't have any experience of dialysis treatment before this study
* Prevalent peritoneal dialysis(PD) patients who are getting peritoneal dialysis treatment more than 6 months
* Prevalent hemodialysis (HD) patients who are getting haemodialysis treatment more than 6 months
* The subjects who are eligible for 1 year follow up
* Written informed consent before any trial related activities
* Eligible patients to complete questionnaire

Exclusion Criteria:

* Prognosis for survival less than 3 months
* Kidney transplantation less than 15 months
* Ineligible patients for questionnaire
* Any malignancies and ascites
* Any condition which could interfere with the patient's ability to comply with the study protocol
* Ineligible to measure BCM

  1. pacemaker, defibrillator
  2. pregnancy or lactation period
  3. amputation
  4. artificial joint

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Incident PD patients group : 250 subjects, First treatment for ESRD by any peritoneal dialysis modality within 30 days prior to or following enrollment (patients may be enrolled prior to commencing first treatment if there is clear indication that the treatment modality is CAPD or APD and they consent in advance to enter the study) and patients who don't have any experience of dialysis treatment before this study
  2. Prevalent PD patients : 250 subjects, Prevalent peritoneal dialysis(PD) patients who are under peritoneal dialysis treatment more than 6 months
  3. Prevalent HD patients : 250 subjects, Prevalent hemodialysis(HD) patients who are under hemodialysis treatment more than 6 months
Sampling Method: Non-Probability Sample
Enrollment: 1068 (Actual)
Dates: Start 2010-08; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yongsoo Kim, M.D., Ph.D., Principal Investigator — Division of nephrology, The Catholic University of Korea College of Medicine
Locations (1):
- Seoul St. Mary's Hospital, Seoul, Seocho-gu, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1. Date of the recruitment period : From October 10, 2010 to April 3, 2013
  2. Types of location : At the general hospitals
Groups:
- Incident Peritoneal Dialysis(PD) Patients: First treatment for end stage of renal disease (ESRD) by any peritoneal dialysis modality within 30 days prior to or following enrollment (patients may be enrolled prior to commencing first treatment if there is clear indication that the treatment modality is continuous ambulatory peritoneal dialysis (CAPD) or automated peritoneal dialysis (APD) and they consent in advance to enter the study) and patients who don't have any experience of dialysis treatment before this study
- Prevalent Peritoneal Dialysis (PD) Patients: Prevalent peritoneal dialysis(PD) patients who are under peritoneal dialysis treatment more than 6 months
- Prevalent Hemodialysis (HD) Patients: Prevalent hemodialysis(HD) patients who are under hemodialysis treatment more than 6 months
Period: Overall Study
Arm/Group | Incident Peritoneal Dialysis(PD) Patients | Prevalent Peritoneal Dialysis (PD) Patients | Prevalent Hemodialysis (HD) Patients
Started | 349 (5 subjects had been excluded due to protocol violation and then data of the rest were anlayzed.) | 359 | 367 (2 subjects had been excluded due to protocol violation and then data of the rest were anlayzed.)
Completed | 347 | 359 | 367
Not Completed | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Incident PD Patients: First treatment for end stage of renal disease (ESRD) by any peritoneal dialysis modality within 30 days prior to or following enrollment (patients may be enrolled prior to commencing first treatment if there is clear indication that the treatment modality is continuous ambulatory peritoneal dia;ysis (CAPD) or automated peritoneal dialysis (APD) and they consent in advance to enter the study) and patients who don't have any experience of dialysis treatment before this study
- Total: Total of all reporting groups
Arm/Group | Incident PD Patients | Prevalent PD Patients | Prevalent HD Patients | Total
Number analyzed (Participants) | 349 | 359 | 367 | 1075
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 279 | 285 | 297 | 861
  >=65 years | 70 | 74 | 70 | 214
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.7 (11.6) | 51.9 (11.6) | 51.0 (11.5) | 51.5 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 209 | 180 | 189 | 578
  Male | 140 | 179 | 178 | 497

OUTCOME MEASURES:

1. Primary Outcome: Change of Kidney Disease Quality of Life Short Form 1.3 (KDQOL SF 1.3) Score and Beck Depression Inventory(BDI) Score From Visit 1 Period
Description: Health-related quality of life (HRQOL) is assessed via KDQOL SF 1.3 and depression is assessed via BDI at the visit 1 and Visit 2 period.
  KDQOL SF 1.3 and BDI are validated questionnaires to assess HRQOL and depression, respectively.
  Visit 2 period is followed 12 months after Visit 1 period. The outcome measure is the difference in averaged scores between Visit 1 and Visit 2; It is calculated as (Score at visit 2 - Score at visit 1).
  HRQOL is assessed by three components; physical health score, mental health score and kidney disease health score.
  Physical health score, mental health score and kidney disease health score are averaged scores of subscales.
  The range of each score and each subscale are 0 - 100, and higher values indicate better HRQOL status.
  The BDI score is a summed score of each component of BDI questionnaire, and the range is 5 to 63. Higher BDI scores are considered to represent more severe depression symptoms.
Time Frame: Visit 1(zero month) and Visit 2 (12 months after Visit 1)
Population: 5 subjects in Incident PD patients and 2 subjects in Prevalent HD patients are excluded due to protocol violation.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Incident PD Patients: First treatment for end stage of renal disease (ESRD) by any peritoneal dialysis modality within 30 days prior to or following enrollment (patients may be enrolled prior to commencing first treatment if there is clear indication that the treatment modality is continuous ambulatory peritoneal dialysis (CAPD) or automated peritoneal dialysis (APD) and they consent in advance to enter the study) and patients who don't have any experience of dialysis treatment before this study
Arm/Group | Incident PD Patients | Prevalent PD Patients | Prevalent HD Patients
Number analyzed (Participants) | 347 | 359 | 367
units on a scale
  Change in Physical health score | 1.22 (19.53) | -1.50 (17.95) | 1.62 (17.44)
  Change in Mental health score | 0.46 (13.39) | -1.27 (12.04) | 0.32 (11.98)
  Change in Kidney disease component score | -1.34 (11.46) | -0.50 (10.03) | -0.95 (10.5)
  Change in BDI score | 1.12 (8.74) | 0.60 (7.90) | -0.08 (7.33)

2. Secondary Outcome: The Association Between Hydration Status and Depression and Quality of Life in Peritoneal Dialysis Patients
Description: Hydration status is checked via BCM(body composition monitor) at Visit 1 and Visit 2 period, as a Overhydration(OH) value.
  Health-related quality of life (HRQOL) is measured via scores of KDQOL SF1.3. Depression was assessed using Beck Depression Inventory (BDI) score. Visit 2 period is followed 12 months after Visit 1 period. HRQOL is assessed by three components; physical health score, mental health score and kidney disease health score.
  Physical health score, mental health score and kidney disease health score are averaged scores of subscales.
  The range of each score and each subscale are 0 - 100, and higher values indicate better HRQOL status.
  The BDI score is a summed score of each component of BDI questionnaire, and the range is 5 to 63. Higher BDI scores are considered to represent more severe depression symptoms.
  The outcome measure is the averaged scores at Visit 1 between the Normohydration group and Overhydration group.
Time Frame: Visit 1(zero month) and Visit 2 (12 months after Visit 1)
Population: PD participants with OH value, HRQOL scores and BDI scores at visit 1 and visit 2 were assessed for this Outcome Measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Normohydration Group: Peritoneal dialysis patients with baseline -2L<OH value <+2L
- Overhydration Group: Peritoneal dialysis patients with baseline OH value >+2L
Arm/Group | Normohydration Group | Overhydration Group
Number analyzed (Participants) | 266 | 215
units on a scale
  Baseline physical health score | 55.5 (16.2) | 51.5 (16.5)
  Baseline mental health score | 50.1 (10.6) | 47.5 (11.1)
  Baseline kidney disease component score | 69.3 (9.6) | 67.0 (9.6)
  Baseline BDI score | 15.1 (9.5) | 16.7 (9.6)
Statistical Analysis 1: Comparison: Normohydration Group vs Overhydration Group; Student's t-test: Comparison of baseline physical health score between Normohydration group and Overhydration group; Test type: Superiority or Other; p = 0.008, t-test, 2 sided
Statistical Analysis 2: Comparison: Normohydration Group vs Overhydration Group; Student's t test: Comparison of baseline mental health score between Normohydration group and Overhydration group; Test type: Superiority or Other; p = 0.008, t-test, 2 sided
Statistical Analysis 3: Comparison: Normohydration Group vs Overhydration Group; Student's t test: Comparison of baseline kidney disease component score between Normohydration group and Overhydration group; Test type: Superiority or Other; p = 0.008, t-test, 2 sided
Statistical Analysis 4: Comparison: Normohydration Group vs Overhydration Group; Student's t test: Comparison of baseline BDI score between Normohydration group and Overhydration group; Test type: Superiority or Other; p = 0.157, t-test, 2 sided

3. Secondary Outcome: The Association Between Hydration Status and Depression and Quality of Life in Hemodialysis Patients
Description: Quality of life was measured via scores of KDQOL SF1.3. Hydration status was measured via body composition monitor as an Overhydration (OH) value Depression was assessed using Beck depression inventory (BDI) score
Time Frame: Visit 1(zero month) and Visit 2 (12 months after Visit 1)
Population: Only prevalent hemodialysis dialysis participants with complete baseline hydration status and scale scores were assessed for this Outcome Measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Normohydration Group: Hemodialysis patients with baseline -2L<OH value <+2L
- Overhydration Group: Hemodialysis patients with baseline OH value >+2L
Arm/Group | Normohydration Group | Overhydration Group
Number analyzed (Participants) | 198 | 159
units on a scale
  Baseline physical health score | 56.28 (15.01) | 51.97 (18.39)
  Baseline mental health score | 49.93 (10.69) | 47.86 (12.29)
  Baseline kidney disease component score | 67.46 (9.34) | 65.51 (10.65)
  Baseline BDI score | 16.06 (8.81) | 16.57 (9.56)

ADVERSE EVENTS:
Time Frame: Visit 1(zero month) and Visit 2 (12 months after Visit 1)
Groups:
- Incident PD Patients: First treatment for ESRD by any peritoneal dialysis modality within 30 days prior to or following enrollment (patients may be enrolled prior to commencing first treatment if there is clear indication that the treatment modality is CAPD or APD and they consent in advance to enter the study) and patients who don't have any experience of dialysis treatment before this study
Arm/Group | Incident PD Patients | Prevalent PD Patients | Prevalent HD Patients
Serious Adverse Events (participants affected / at risk) | 37/349 | 50/359 | 21/367
Other Adverse Events (participants affected / at risk) | 0/349 | 3/359 | 1/367
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Incident PD Patients (N=349) | Prevalent PD Patients (N=359) | Prevalent HD Patients (N=367)
Peritonitis (Infections and infestations) | 19 (19) | 22 (22) | 0 (0)
Death (Cardiac disorders) | 12 (12) | 21 (21) | 13 (13)
Admission (Renal and urinary disorders) | 6 (6) | 7 (7) | 8 (8)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Incident PD Patients (N=349) | Prevalent PD Patients (N=359) | Prevalent HD Patients (N=367)
Kidney transplantation (Surgical and medical procedures) | 0 (0) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No